CLINICAL TRIAL: NCT06115395
Title: Efficacy and Safety of Using Non-invasive Ventilation Assisted Fiber-optic Bronchoscopy
Brief Title: Non-invasive Ventilation Assisted Fiber-optic Bronchoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Walaa Maher Abd El aziz, Principal Investigator Walaa Maher abd El aziz, Head of NIV Ahmed Younis El-sayed, Clinical Professor Amr Abd El-Hamid Moawad and Director Mohamed Ahmed Mansour Affiliation: Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Bronchoscopy with NIV
Record Dates: First submitted 2023-09-09; First posted 2023-11-03 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Lung; Diseases
Keywords: non- invasive ventilation; fiber-optic bronchoscopy.
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: Sample method:
  Method of randomization was stratified random sampling method was adopted to create matched study groups. Patients admitted for bronchoscopy were classified into two categories:
  1. A) Non hypoxemic group.
  2. B) Hypoxemic group.
  3. From each category: 50 patients were selected and allocated randomly in the study groups (either intervention or control group) using lottery method. So, each study group with included 25 patients from each category forming a total of 50 patients in each studies categories.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- (Group 1) 25 (H. NIV): Hypoxemic patients{hypoxemic NIV group} (Active Comparator): who will undergo fiber-optic bronchoscopy under non- invasive ventilation and conventional oxygen therapy
  Interventions: Device: non- invasive ventilator; Device: fiber-optic bronchoscopy
- (Group 2) 25 (H. conv.): Hypoxemic patients{hypoxemic conventional group } (Active Comparator): who will undergo conventional fiber-optic bronchoscopy under conventional oxygen therapy without non- invasive ventilation
  Interventions: Device: fiber-optic bronchoscopy
- (Group 3) 25 (N.H.NIV): Non- hypoxemic patients{non-hypoxemic NIV group} (Active Comparator): who will undergo fiber-optic bronchoscopy under non- invasive ventilation and conventional oxygen therapy
  Interventions: Device: non- invasive ventilator; Device: fiber-optic bronchoscopy
- (Group 4) 25(N.H. conv.): Non- hypoxemic patients{non-hypoxemic conventional group} (Active Comparator): who will undergo conventional fiber-optic bronchoscopy under conventional oxygen therapy without non- invasive ventilation
  Interventions: Device: fiber-optic bronchoscopy

INTERVENTIONS:
Device: non- invasive ventilator — Group 1 (hypoexemic patient who will undergo bronchoscopy under non- invasive ventilation{NIV} and conventional o2 therapy) will be on NIV half an hour prior and throughout the bronchoscopic sampling and after the procedure until reach the baseline criteria
  Other Names: fiber-optic bronchoscopy; conventional oxygen therapy
  Arms: (Group 1) 25 (H. NIV): Hypoxemic patients{hypoxemic NIV group}; (Group 3) 25 (N.H.NIV): Non- hypoxemic patients{non-hypoxemic NIV group}
Device: fiber-optic bronchoscopy — Group 2 (hypoxemic patients who will undergo conventional bronchoscopy under conventional o2 therapy without NIV ) will be on conventional oxygen therapy half an hour prior and throughout the bronchoscopic sampling and after the procedure until reach the baseline criteria
  Other Names: conventional bronchoscopy under oxygen therapy; conventional oxygen therapy
Device: non- invasive ventilator — Group 3 (non- hypoxemic patients who will undergo bronchoscopy under non- invasive ventilation{NIV} and conventional o2 therapy) will be on NIV throughout the bronchoscopic sampling and after the procedure until reach the baseline criteria
  Other Names: fiber-optic bronchoscopy; conventional oxygen therapy
  Arms: (Group 1) 25 (H. NIV): Hypoxemic patients{hypoxemic NIV group}; (Group 3) 25 (N.H.NIV): Non- hypoxemic patients{non-hypoxemic NIV group}
Device: fiber-optic bronchoscopy — Group 4 (non- hypoxemic patients who will undergo conventional bronchoscopy without non- invasive ventilation{NIV) will be on conventional oxygen therapy throughout the bronchoscopic sampling and after the procedure until reach the baseline criteria
  Other Names: conventional bronchoscopy under oxygen therapy; conventional oxygen therapy

SUMMARY:
The purpose of this study is the evaluation of using bi-level positive airway pressure ventilation in candidates for fiber-optic bronchoscopy regarding benefits and drawbacks.

DETAILED DESCRIPTION:
In this study patients who will be candidate for fiber-optic bronchoscopy for diagnostic or therapeutic reasons will be evaluated by the Chest Medicine Department, Mansoura University Hospitals. All patients will be subjected to full history taking, full examination, routine laboratory investigations, arterial blood gases (ABG), chest X-ray, chest computed tomography (CT). Non-invasive ventilation: Group 1 (hypoexemic patient who will undergo bronchoscopy under non- invasive ventilation{NIV}) will be on NIV half an hour prior and throughout the bronchoscopic sampling and after the procedure until reach the baseline criteria, Group 2 (hypoxemic patients who will undergo conventional bronchoscopy ) will be on conventional oxygen therapy half an hour prior and throughout the bronchoscopic sampling and after the procedure until reach the baseline criteria, Group 3 (non- hypoxemic patients who will undergo conventional bronchoscopy ) will be on NIV throughout the bronchoscopic sampling and after the procedure until reach the baseline criteria, Group 4 (non- hypoxemic patients who will undergo conventional bronchoscopy) will be on conventional oxygen therapy throughout the bronchoscopic sampling and after the procedure until reach the baseline criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients who admitted to the pulmonology ward or intensive care unit with any (diagnostic and/or therapeutic) bronchoscopy indication.

  1. Age 18 years or more.
  2. Patients accepted to participate in the study.

Exclusion Criteria:

* Patients with:

  1. Cardiac or respiratory arrest.
  2. Impaired consciousness or confusion.
  3. Type II respiratory failure.
  4. Hemodynamic instability.
  5. Inability to cooperate or to protect the airway.
  6. Vomiting, bowel obstruction, recent upper gastrointestinal tract surgery and esophageal injury.
  7. Patients refusing participation in the study.
  8. Patients unfit for NIV and or NIV mask.
  9. Intubation and or invasive ventilation candidates.
  10. Presence of contraindications for bronchoscopy procedure such as insufficient platelet number or coagulopathy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-25 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the changes in oxygen saturation, heart rate, respiratory rate, blood pressure, dyspnea score and arterial blood gases in bronchoscopy procedure | 4 years
  Evaluate changes and when to reach base line in each of 1- (SPO2) by pulse oximeter in (percentage %) at base line, 15 minute before, during and immediately after bronchoscopy.
  2-heart rate in (beat/minute) at base line, 15 minute before, during and immediately after bronchoscopy.
  3-respiratory rate in (cycle/minute) at base line, 15 minute before, during and immediately after bronchoscopy.
  4-mean arterial blood pressure in {millimeter/mercury mm/Hg)} at base line, 15 minute before, during and immediately after bronchoscopy.
  5-dyspnea score in {grade 0-3 according to: (mMRC)} 15 minute before and immediately after bronchoscopy.
  arterial blood gases (PH, Paco2 in {millimeter/mercury (mm/Hg)}, Pao2 in {millimeter/mercury (mm/Hg)},Spo2 (percentage %) andHco3 in {millimol (mmol/l)} before and after bronchoscopy.
  To show effects of using NIV and conventional o2 therapy and using of conventional o2 therapy alone on these parameters in the studied patients in bronchoscopy.

SECONDARY OUTCOMES:
Fiber-optic bronchoscopy complications | 4 years
  The need for intubation, if it occurs within two to eight hours of bronchoscopy, it was considered as a complication possibly related to bronchoscopy. This time span was adopted from previous studies (Hilbertet et al., 2001). Also the existence of complications as hemorrhage, pneumothorax, hypotension, arrhythmia) that occurred during bronchoscopy and in the first 24 hours following bronchoscopy, which could possibly be related to the procedure (Schönhofer et al., 2008).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El sayed, MD, Study Chair — Mansoura University; Amr Moawad, MD, Study Director — Mansoura University; Mohamed Mansour, MD, Study Director — Mansoura University
Locations (1):
- Walaa Maher Abd ElAziz,, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Biswas A, Mehta H, Sriram P. Diagnostic Yield of the Virtual Bronchoscopic Navigation System Guided Sampling of Peripheral Lung Lesions using Ultrathin Bronchoscope and Protected Bronchial Brush. Turk Thorac J. 2019; 01; 20(1):6-11. 2. Campos JH. Fiberoptic bronchoscopy guidelines for the anesthesiologist. Revista Mexicana de Anestesiología. 2011; 31: S264-9. 3. Hilbert G, Gruson D, Vargas F, Valentino R, Favier JC, Portel L, et al. Bronchoscopy with bronchoalveolar lavage via the laryngeal mask airway in high-risk hypoxemic immunosuppressed patients. Crit Care Med. 2001; 29: 249-255. 4. Schönhofer B, Kuhlen R, Neumann P, et al. Non-invasive ventilation as treatment for acute respiratory insufficiency. Essentials from the new S3 guidelines. Anaesthesist. 2008; 57: 1091-102.